CLINICAL TRIAL: NCT00411723
Title: Phase 1 Safety Study of RTL1000 (Recombinant T Cell Receptor Ligand) in Subjects With Multiple Sclerosis
Brief Title: Safety Study of RTL1000 (Recombinant T Cell Receptor Ligand) in Subjects With Multiple Sclerosis
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Artielle ImmunoTherapeutics (Industry)
Responsible Party: Andrew S. Goldstein, Artielle ImmunoTherapeutics, Inc.
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RTL1000-1.0001
Record Dates: First submitted 2006-12-12; First posted 2006-12-14 (Estimated); Last update posted 2009-02-20 (Estimated); Status verified 2009-02

CONDITIONS: Multiple Sclerosis, Chronic Progressive; Multiple Sclerosis, Relapsing-Remitting
Keywords: multiple sclerosis, chronic-progressive, relapsing-remitting
MeSH Terms: conditions — Multiple Sclerosis, Chronic Progressive; Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: RTL1000 (recombinant T cell receptor ligand)
- 2 (Placebo Comparator)
  Interventions: Drug: RTL1000 Placebo

INTERVENTIONS:
Drug: RTL1000 (recombinant T cell receptor ligand) — Dosage form: IV infusion. Dosage: Single dose @ 2, 6, 20, 60, 100 or 200mg. Duration: 1 - 2 hours.
  Arms: 1
Drug: RTL1000 Placebo — Dosage form: IV infusion. Dosage: Same volume as Experimental. Frequency: Single dose. Duration: 1 - 2 hours.
  Arms: 2

SUMMARY:
RTL1000 is a new agent that has not been previously tested in humans. It is thought that RTL may specifically control the abnormal immune response or attack against the insulation on the nerves that occurs in multiple sclerosis.

The purpose of this study is to evaluate the possible side effects of a single intravenous dose of RTL1000 in subjects with multiple sclerosis. Some subjects will also be asked to participate in one or both of two substudies, one to test blood samples to see how the body's immune system responds after administration of RTL1000, and the other to test blood samples to see how the body absorbs and eliminates the RTL1000.

DETAILED DESCRIPTION:
This is a double-blind, placebo-controlled treatment protocol with up to six treatment cohorts, each of which receives a single intravenous infusion of an escalating dose of RTL1000. Each dosing group will have six subjects: two who will receive a single dose of placebo and four who will receive a single dose of RTL1000. Subjects are observed in the hospital during the infusion and for 24 hours afterward, and are then followed weekly for 28 days and at 1 and 2 months post-infusion to evaluate safety parameters.

Objectives of the study are to evaluate the safety profile of a single dose of RTL1000 administered by intravenous infusion, to evaluate the pharmacokinetic profile of RTL1000 in a subset of subjects, and to evaluate the feasibility of assessing immunologic parameters in a subset of subjects.

Endpoints include vital signs, electrocardiogram and physical examination results, adverse events, and serious adverse events and safety laboratory parameters (e.g., clinical chemistries and hematology values). Disease parameters, such as neurological findings, expanded disability status scale (EDSS), 25-ft timed walk, 9-hole peg test, and magnetic resonance imaging (MRI) will be measured to ensure that study treatment does not make disease worse. Subjects will also be tested at the beginning and end of the study for antibodies to the drug and its components.

ELIGIBILITY:
A specific blood cell type called HLA-DR2 may be required in order for RTL1000 to work. For that reason, all subjects will be tested for HLA-DR2 and only those subjects who test positive (about 50%) will undergo further tests to determine if they meet inclusion and exclusion criteria.

Inclusion criteria:

* Fulfill McDonald criteria for multiple sclerosis
* Confirmed diagnosis of chronic progressive or relapsing-remitting multiple sclerosis
* EDSS score of 0.0 to 6.5
* No clinical exacerbations within the 8 weeks before administration of RTL1000
* HLA-DR2 positive, as confirmed by study reference laboratory
* Negative serum pregnancy test within 7 days of administration of RTL1000 and negative urine pregnancy test on Day 0 for all women of childbearing potential
* Agreement of sexually active men and women of childbearing potential to practice a medically-approved form of contraception
* Capable of and willing to provide written informed consent

Exclusion Criteria:

* Exposure to alemtuzumab or dacluzimab any time in the 6 months before administration of RTL1000
* Exposure to natalizumab or other drugs targeting alpha-4 integrin in the 6 months before RTL1000 administration or more than 3 doses of natalizumab or these drugs at any time.
* Any prior exposure to RTL1000
* Exposure to other MS disease-modifying drugs (e.g., recombinant interferon beta and glatiramer acetate), immunosuppressant agents, or systemic corticosteroids (other than replacement doses) within the 4 weeks prior to RTL1000 administration
* Exposure to chemotherapeutic immunosuppressants, including azathioprine, mycophenolate mofetil, methotrexate, cladribine, mitoxantrone, or cyclophosphamide, during the six months prior to administration of RTL1000
* Total lymphoid irradiation or bone marrow transplantation at any time
* Known or suspected allergy to gadolinium
* Contraindication to MRI (e.g., subject has a pacemaker or other contraindicated implanted metal devices or has claustrophobia that cannot be medically managed)
* Clinically significant abnormalities in laboratory findings for hematologic, hepatic, and renal function at screening.
* Significant medical diseases or conditions, including poorly controlled hypertension, cardiovascular disease, inflammatory disorders, immunodeficiency (e.g., HIV infection), renal failure, liver dysfunction, cancer (except treated basal cell carcinoma), or active infection.
* History of, or current, psychiatric illness likely to interfere with ability to comply with protocol requirements or give informed consent
* History of alcohol or drug abuse likely to interfere with ability to comply with protocol requirements
* Pregnancy or lactation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2006-12; Primary Completion 2009-02 (Actual); Study Completion 2009-05 (Estimated)

PRIMARY OUTCOMES:
Adverse events, safety, laboratory parameters, vital signs, ECG and physical exam results. Disease parameters (neurologic exam, EDSS, 25 foot timed walk, 9-hole PEG test, MRI). Antibodies to drug. | Day 28

CONTACTS AND LOCATIONS:
Overall Officials: Jana Preiningerova, M.D., Principal Investigator — Yale Center for MS Treatment and Research; David Mattson, M.D., Ph.D., Principal Investigator — University of Indiana, Department of Neurology; Sharon Lynch, M.D., Principal Investigator — University of Kansas Medical Center, Landon Center on Aging; Christopher Bever, Jr., M.D., M.B.A., Principal Investigator — University of Maryland, Baltimore; Theodore R Brown, M.D., Principal Investigator — MS Center at Evergreen; Vijayshree Yadav, M.D., Principal Investigator — MS Center of Oregon Health and Science University
Locations (6):
- United States (6):
  - Yale Center for MS Treatment and Research, New Haven, Connecticut
  - Indiana University, Dept. of Neurology, Indianapolis, Indiana
  - University of Kansas Medical Center, Landon Center on Aging, Kansas City, Kansas
  - University of Maryland School of Medicine, Baltimore, Maryland
  - MS Center of Oregon Health & Science University, Portland, Oregon
  - MS Center at Evergreen, Kirkland, Washington